CLINICAL TRIAL: NCT00752167
Title: Diagnosis of EIB and Asthma in NCAA Division I Athletes
Brief Title: Diagnosis of Exercise-induced Bronchospasm (EIB) and Asthma in National Collegiate Athletic Association (NCAA) Division I Athletes
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: GSK 110189
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2008-09

CONDITIONS: Exercise Induced Bronchospasm, Asthma
Keywords: exercise induced bronchospasm; asthma; athlete; sports; eucapnic voluntary hyperventilation; albuterol
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: all Division I athletes, male and female, at the University of Arizona that are currently being treated for either EIB or asthma by review of preparticipation physical forms or identified by the medical staff
- Control: control athletes (ie, not currently being treated for either EIB or asthma by review of preparticipation physical forms or identified by the medical staff and/or not currently using asthma medications) from the same sport

SUMMARY:
We hypothesize that exercise-induced bronchospasm (EIB) at the NCAA Division I collegiate level is over diagnosed, while poorly controlled asthma resulting in exercise-related symptoms in this same population may be under diagnosed, being erroneously attributed to EIB. This project will test individuals self-identified as having exercise induced bronchospasm or asthma, as well as gender-matched controls from the same sport, with eucapnic voluntary hyperventilation to assess for the presence of EIB or asthma. By making the correct diagnosis, improved health outcomes may be achieved and athletic performance may be enhanced.

DETAILED DESCRIPTION:
We plan to identify all Division I athletes, male and female, at the University of Arizona that are currently being treated for either EIB or asthma by review of preparticipation physical forms or identified by the medical staff. In addition, athletes that were prescribed inhalers through Campus Health Services will be identified through review of electronic pharmacy records. Each athlete identified will be matched with two control athletes (ie, not currently using asthma medications) from the same sport. Subjects will be tested for EIB using eucapnic voluntary hyperventilation, the gold standard for making this diagnosis.

Subject Recruitment Potential subjects will be identified as described above. Subjects will be approached by one of the co-investigators, the study explained and an opportunity to review the consent form and ask question provided. Subjects who consent will then be scheduled for testing.

Questionnaire Subjects, once enrolled, will be asked to complete a 27 item questionnaire including questions about prior history and treatment of asthma, as well as history of respiratory symptoms. In addition, subjects will be asked to complete the Asthma Control Test (ACT).

EVH and Spirometric Testing All subjects will undergo baseline assessment of lung function using the KoKo Legend Portable Spirometer. The subjects will then undergo eucapnic voluntary hyperventilation testing. EVH testing will require the subject to hyperventilate dry air containing 5% carbon dioxide at room temperature for six minutes at a target ventilation of 30 times the subject's forced expiratory volume in one second (FEV1). The EVH test will be considered positive if a fall in FEV1 of 10% or more from baseline is recorded after a 6 minute period of hyperpnea. To overcome the problem of any post-test respiratory muscle fatigue, the FEV1 will be recorded at least three minutes after challenge and then repeated at three-minute intervals through 21 minutes.

Spirometry will be carried out according to American Thoracic Society standards. Both absolute and percent-predicted spirometric values will be recorded. Predicted values will be calculated from validated, published, race-specific regression equations. (Hankinson, et al. Spirometric reference values values from a sample of the general US population. Am J Respir Crit Care Med 1999; 159:179-187.) Asian-American athletes will be evaluated using norms for whites.

To provide the optimal test circumstances, some medications will be withheld for 8 to 96 hours before the bronchial provocation test: no short-acting bronchodilators, sodium cromoglycate, nedocromil sodium, or ipratropium bromide for 8 hours; no long-acting bronchodilators or antihistamines for 48 hours; no leukotriene antagonists for four days. Steroids should not be inhaled on the day of the test. No caffeine should be taken on the morning of the test. Vigorous exercise will be avoided for at least four hours prior to the start of the test as well as any exercise on the day of testing. Subjects will be scheduled for testing to allow at least 6-8 hours to elapse between previous vigorous activity and testing.

Exhaled Nitric Oxide (eNO) Measurement

Measurement of eNO will be obtained prior to measurement of pre-EVH spirometry. Exhaled NO will be measured employing a technique modified after Silkoff et al (1997) and following American Thoracic Society guidelines for eNO assessment (American Thoracic Society, 1999). In brief, this technique utilizes a resistive device that provides a constant low expiratory flow rate and ensures vellum closure. The combination of vellum closure and low flow rates, specifically 50 ml/s, assures accurate measurement of specific pulmonary derived eNO, while excluding potential contamination by nasal and paranasal sinuses NO (which can be a large source of eNO). Nitric oxide concentrations will be measured using a rapid-response chemiluminescent analyzer (NIOX™ System, Aerocrine, Sweden), which has a response time of < 700 ms for 10-90% full scale. The Food and Drug Administration has approved this device for clinical application in asthma management. The measurement circuit will consist of a mouthpiece-filter connected to a resistor/flow meter and collection bag. The participant will inhale to total lung capacity (TLC), insert the mouthpiece, and then immediately exhale slowly. During expiration, the participant will attempt to maintain a target flow of 50 ml/sec. The target period of exhalation time will be 10 seconds. However, for participants that are not able to perform the 10 second exhalation, the time requirements may be decreased to 6 seconds. Dietary history by recall for the 4-6 hours prior to testing will be obtained to screen for dietary sources of NO.

Data Collection Spirometric values and quality control measures for EVH testing will be recorded on forms specifically designed for this purpose and, for spirometry, already in use in the Pediatric Pulmonary Function Laboratory. Data will entered into a computer spreadsheet and double-checked by a second person to assure accuracy. It will then be transferred to a statistical package (STATA) for subsequent analysis.

Data Analysis For this observational study summative and descriptive statistics will be carried out. If opportunities for comparative analysis are identified, parametric and nonparametric analysis will be carried out as appropriate.

A fall occurring early in the post-EVH period, especially in conjunction with documented pre-exercise elevation in eNO, will be taken as being more suggestive of poorly controlled asthma, while a fall 9-12 minutes after EVH, especially in the absence of an elevated eNO, will be interpreted as being more indicative of true EIB.

ELIGIBILITY:
Inclusion Criteria:

* varsity athlete
* ability and willingness to give written informed consent

Exclusion Criteria:

* inability to give written informed consent
* unwillingness to perform spirometry or eucapnic voluntary hyperventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NCAA Varsity Division I athletes attending the University of Arizona
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 following eucapnic voluntary hyperventilation | 3-21 minutes

SECONDARY OUTCOMES:
Protection from fall in FEV1 following eucapnic voluntary hyperventilation by preadministration of albuterol | 3-21 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David Millward, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Millward D, Paul S, Brown M, Porter D, Stilson M, Cohen R, Olvey E, Hagan J. The diagnosis of asthma and exercise-induced bronchospasm in division I athletes. Clin J Sport Med. 2009 Nov;19(6):482-6. doi: 10.1097/JSM.0b013e3181bcde2c. PMID 19898076